CLINICAL TRIAL: NCT00567710
Title: A Six-week, Randomized, Double-blind, Placebo-controlled, Parallel Group, Multi-center, Phase II Study to Determine the Efficacy, Tolerability and Safety of Low and High Non-overlapping Dose Ranges of BL-1020 Compared to Placebo and Risperidone
Brief Title: A Six-week, Randomized, Double-blind, Placebo-controlled, Parallel Group, Multi-center, Phase II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: BioLineRx, Drug development Company
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BL - 1020 IIb; BL - 1020 IIb
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — perphenazine GABA ester; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- I (Experimental): BL - 1020 lowdose
  Interventions: Drug: BL - 1020
- II (Experimental): BL 1020 high dose
  Interventions: Drug: BL - 1020
- III (Placebo Comparator)
  Interventions: Drug: Placebo
- IV (Active Comparator): Risperidone
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: BL - 1020 — 10 mg/day
  Arms: I
Drug: BL - 1020 — BL 1020 20-30 mg/day
  Arms: II
Drug: Placebo — Capsules
  Arms: III
Drug: Risperidone — Capsules
  Arms: IV

SUMMARY:
This is a prospective, six-week, randomized, double blind, placebo-controlled, multi-center study in patients with schizophrenia who are experiencing an acute exacerbation of psychosis.

DETAILED DESCRIPTION:
This study consists of a 5- to 14-day screening period to include antipsychotic medication washout, followed by a six-week double blind treatment period. Patients completing the 6-week treatment period may continue double-blind treatment in an optional extension period of at least 6 weeks' duration. Patients randomized to placebo during the initial 6-week period will be randomized to BL-1020 low or high dose during the extension treatment period. Approximately 40 study centers in four countries will participate.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female, 18-65 years of age, inclusive.
* If female, the patient must be post-menopausal, or if fecund, must be abstinent or practicing an established method of birth control such as hormonal preparations (e.g., oral contraceptive tablets, hormonal implant device, hormone patch, or injectable contraceptive), or intrauterine device [IUD], for at least two months prior to screening, and in addition must use a barrier method, e.g., condom, diaphragm, contraceptive foam.
* Patient is willing and able to provide informed consent, after the nature of the study has been fully explained.
* Patient is an inpatient or outpatient who has a current DSM-IV-TR diagnosis of schizophrenia, as confirmed by the MINI-Plus.
* Patient must be experiencing an acute exacerbation of psychosis, with a baseline (Study Day 0) total score on the PANSS greater than '70'.
* Patient must have a score of '4' ("moderate") or more at baseline on two of the following four PANSS items: delusions, hallucinatory behaviors, conceptual disorganization or suspiciousness/persecution, where at least one of the two items must be either delusions or hallucinatory behaviors, and the total score on the four items must be greater than '17'.
* Patient must be experiencing an acute exacerbation of psychosis with a total score on the CGI-S of '4' ("moderate") or greater at baseline.
* Patient is willing to be hospitalized at screening, and willing to remain in the hospital at least 14 days after baseline (through Study Day 14) as clinically indicated, and must be willing to comply with all study related evaluations and procedures through Study Day 42.
* Patient has a caregiver or an identified responsible person (e.g., family member, social worker, nurse) who will support him/her to ensure compliance with the treatment and outpatient visits.
* Patient is willing to comply with not taking any prohibited medications during participation in the study.

Exclusion Criteria:

* The presence of any of the following will exclude a patient from study enrolment:

General

* Patient is unwilling or unable to provide informed consent.
* Patient is unwilling or unable, in the opinion of the Investigator, to comply with study instructions.
* If female, patient is pregnant, breast-feeding, has a positive urine pregnancy test at screening or baseline, or is of reproductive capacity and is unwilling to comply with accepted contraceptive methods during the study, ie, not using an oral contraceptive, hormonal patch or implant, injectable contraceptive or IUD, in combination with a barrier method (see Inclusion Criterion #2).
* Patient has made a plasma or blood donation within 14 days prior to the screening visit.
* Patient has participated in a prior clinical study of BL-1020 or any of its excipients, and/or has received an investigational drug within thirty days prior to screening.
* Patient is judged by the PI to be inappropriate for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
to evaluate the safety and tolerability of two dose ranges | 6 weeks

SECONDARY OUTCOMES:
to evaluate the efficacy of two dose ranges | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yona Geffen, Ph.D, Study Director — BioLineRx, Ltd.
Locations (1):
- Mary ann Knisevich, Irving, Texas, United States

REFERENCES:
- [Derived] Geffen Y, Keefe R, Rabinowitz J, Anand R, Davidson M. Bl-1020, a new gamma-aminobutyric acid-enhanced antipsychotic: results of 6-week, randomized, double-blind, controlled, efficacy and safety study. J Clin Psychiatry. 2012 Sep;73(9):e1168-74. doi: 10.4088/JCP.12m07642. PMID 23059159